CLINICAL TRIAL: NCT03209089
Title: A Non-Interventional Study on Type 2 Diabetes Mellitus Patient's Characteristics and Management by General Practitioners and Endocrinologists in the Russian Population (THESEUS)
Brief Title: Type 2 Diabetes Mellitus Patients' Characteristics and Management by General Practitioners and Endocrinologists
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00037
Record Dates: First submitted 2017-06-19; First posted 2017-07-06 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-centre observational, ambispective study, which will retrospectively and prospectively collect clinical variables and socio-demographic data from medical records of patients with type 2 diabetes mellitus (T2DM) initiated with dapagliflozin by general practitioners (GPs) and endocrinologists in real-life setting. It is anticipated that patient recruitment will last 8 months (from Q3 2017 to Q1 2018) and each patient will be followed during the second visit 6±3 months later after the first visit. There are 2 time points:

* Baseline data: baseline data are defined as data available within 3 months prior to the first dose of dapagliflozin. In case of presence of multiple data values within baseline period the most recent pre-dose value will be selected
* Follow-up data: any post-baseline data will be considered as follow-up but the primary analysis will be focused on data available at 6±3 months after the first visit. In case of discontinuation dapagliflozin, data will be collected at routine visit within 3-month time frame after the last dose

DETAILED DESCRIPTION:
Study design:

This is a multi-centre observational, ambispective study, which will retrospectively and prospectively collect clinical variables and socio-demographic data from medical records of patients with T2DM initiated with dapagliflozin by GPs and endocrinologists in real-life setting.

Only patients, who provide written consent to participate in the study will be enrolled into this study. All patients will be unique with no overlap between endocrinologists and GPs. All consecutive patients managed by GPs or endocrinologists who meet inclusion criteria will be included. All GPs and endocrinologists, who manage T2DM on sites, will be participating investigators.

Patients will undergo clinical assessment and receive the standard medical care as usual determined by the treating doctor based on their clinical judgement and national guidelines. Patients will not receive experimental treatment as a consequence of their participation in the observational study.

It is anticipated that patient recruitment will last for 8 months (from Q3 2017 to Q1 2018) and each patient will be followed during the second visit 6±3 months later after the first visit.

There are 2 time points:

* Baseline data: baseline data are defined as data available within 3 months prior to the first dose of dapagliflozin. In case of presence of multiple data values within baseline period the most recent pre-dose value will be selected
* Follow-up data: any post-baseline data will be considered as follow-up but the primary analysis will be focused on data available at 6±3 months after the first visit. In case of discontinuation dapagliflozin, data will be collected at routine visit within 3-month time frame after the last dose.

Data Source(s):

Baseline data will be collected during Visit 1 from the T2DM patient medical records, including disease history of patient, and during follow-up data during Visit 2 (after 6±3 months from Visit 1).

Study Population:

It is planned to include 900 male and female T2DM outpatients 18 years and older, who were managed by GPs or endocrinologists in 45 outpatient sites.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older;
* Established diagnosis of T2DM (ICD-10 code E11.2-E11.9)
* The current treatment with dapagliflozin prescribed at least 1 month before the FSI;
* Written voluntary informed consent has been provided
* Management in outpatient setting.

Exclusion Criteria:

* Type 1 diabetes
* Current participation in a clinical trial
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).
* Presence of serious/severe co-morbidities in the opinion of the investigator, which may limit treatment approach as usual.
* Treatment with drugs affecting glucose homeostasis (e.g., systemic glucocorticosteroids) within 3 months before to the 1st Visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 900 male and female T2DM outpatients, who were managed by GPs or endocrinologists in 45 outpatient sites.
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Demographic parameters before dapagliflozin initiation in T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  mean age
demographic characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  age distribution
demographic characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  gender distribution
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  mean duration of T2DM
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  HbA1c (mean and distribution)
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Weight (mean)
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  SBP (mean and distribution)
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  DBP (mean and distribution)
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Proportion of T2DM patients with diabetic complications
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Proportion of patients with T2DM treatment intensification during 3 months before inclusion in the study
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Proportion of patients with different treatment regimen
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Proportion of patients on treatment with different classes of antidiabetic therapy
clinical characteristics of T2DM patients managed by GPs | 3 months before dapagliflozin initiation
  Proportion of patients on different classes of concomitant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Bulatov, MD, PhD, Study Director — AstraZeneca Russia
Locations (20):
- Russia (20):
  - Research Site, Belgorod Region, Shebekino, Russian Federation
  - Research Site, Belgorod Region, Volokonovsky R-n, P. Volokonovka, Russian Federation
  - Research Site, Gis-Khrustalny, Russian Federation
  - Research Site, Izhevsk, Russian Federation
  - Research Site, Kazan', Russian Federation
  - Research Site, Lipetsk, Russian Federation
  - Research Site, N. Novgorod Region, Russian Federation
  - Research Site, Nizhny Novgorod, Russian Federation
  - Research Site, Novomoskovsk, Russian Federation
  - Research Site, Novosibirsk, Russian Federation
  - Research Site, Perm, Russian Federation
  - Research Site, Ryazan, Russian Federation
  - Research Site, Saint Petersburg, Russian Federation
  - Research Site, Samara, Russian Federation
  - Research Site, Tambov Region, Russian Federation
  - Research Site, Volzhsk, Russian Federation
  - Research Site, Voronezh, Russian Federation
  - Research Site, Voronezh Region, Novovoronezh, Russian Federation
  - Research Site, Yaroslavl, Russian Federation
  - Research Site, Yoshkar-Ola, Russian Federation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D1690R00037 Study Report Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00037&attachmentIdentifier=a97b4607-27ff-40cf-8480-559120caac2c&fileName=D1690R00037StudyReportSynopsis.pdf&versionIdentifier=